CLINICAL TRIAL: NCT01270880
Title: A Phase II Trial of STA-9090 in Patients With Metastatic Castration-Resistant Prostate Cancer (CRPC) Pretreated With Docetaxel Based Chemotherapy
Brief Title: Hsp90 Inhibitor STA-9090 in Treating Patients With Metastatic Hormone-Resistant Prostate Cancer Previously Treated With Docetaxel-Based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elisabeth Heath, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-070; NCI-2010-02328 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Results first posted 2015-04-14 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-02

CONDITIONS: Adenocarcinoma of the Prostate; Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — STA 9090; Polymerase Chain Reaction; Enzyme-Linked Immunosorbent Assay; Spectrophotometry; Reverse Transcriptase Polymerase Chain Reaction; Gene Expression Profiling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive Hsp90 inhibitor STA-9090 IV over 1 hour once weekly in weeks 1-3. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Hsp90 inhibitor STA-9090; Other: laboratory biomarker analysis; Genetic: polymerase chain reaction; Other: enzyme-linked immunosorbent assay; Genetic: RNA analysis; Other: spectrophotometry; Genetic: reverse transcriptase-polymerase chain reaction; Genetic: gene expression analysis

INTERVENTIONS:
Drug: Hsp90 inhibitor STA-9090 — Given IV
  Other Names: STA-9090
Other: laboratory biomarker analysis — Correlative studies
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR
Other: enzyme-linked immunosorbent assay — Correlative studies
  Other Names: ELISA
Genetic: RNA analysis — Correlative studies
Other: spectrophotometry — Correlative studies
Genetic: reverse transcriptase-polymerase chain reaction — Correlative studies
  Other Names: RT-PCR
Genetic: gene expression analysis — Correlative studies

SUMMARY:
Hsp90 inhibitor STA-9090 may stop the growth of tumor cells by blocking some of the proteins needed for cell growth. This phase II trial is studying how well Hsp90 inhibitor STA-9090 works in treating patients with metastatic hormone-resistant prostate cancer previously treated with docetaxel-based chemotherapy

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate progression-free survival (PFS) achieved with STA-9090 (Hsp90 inhibitor STA-9090) in men with castration-resistant prostate cancer (CRPC) who have received prior docetaxel based therapy.

SECONDARY OBJECTIVES:

I. To assess the percentage change in prostate-specific antigen (PSA) from baseline to 12 weeks.

II. To assess overall safety and tolerability of STA-9090. III. To evaluate overall survival (OS) outcome in metastatic CRPC who have received prior docetaxel therapy.

IV. To investigate the association of progression-free survival (PFS) and PSA response rate with primary and secondary target markers.

TERTIARY OBJECTIVES:

I. To evaluate potential markers for predicting drug response or efficacy, blood samples will be used to collect the serum and extract messenger ribonucleic acid (mRNA) from mononuclear cells and analyzed by quantitative real-time polymerase chain reaction (PCR) and/or enzyme-linked immunosorbent assay (ELISA).

OUTLINE:

Patients receive Hsp90 inhibitor STA-9090 intravenously (IV) over 1 hour once weekly in weeks 1-3. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of prostate adenocarcinoma with metastasis and objective progression or rising PSA despite androgen deprivation therapy and antiandrogen withdrawal when applicable
* Progression after docetaxel based chemotherapy is needed as follows:
* a) If measurable disease present, then either rising PSA, increase in size of the lesion/s or both should be present
* b) Patients with rising PSA only as progression must demonstrate a rising trend with 2 successive elevations at minimum intervals of 1 week; a minimum PSA of 5 ng/ml, or new areas of bony metastases on bone scan are required for patients with no measurable disease; no minimum PSA requirement for patients with measurable disease
* Patients should have received at least one prior docetaxel based regimen for metastatic disease; no maximum prior therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 2
* Life expectancy of at least 3 months
* Prior radiation therapy or chemotherapy completed at least 28 days prior to enrollment
* All patients must be documented to be castrate with a testosterone level =< 0.5 ng/ml; luteinizing-hormone-releasing hormone (LHRH) agonist therapy must be continued, if required to maintain castrate levels of testosterone; patients must be off antiandrogens for a minimum of 4 weeks for flutamide and 6 weeks for bicalutamide or nilutamide
* Absolute neutrophil count >= 1,500 cells/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 9.0 g/dL
* Serum creatinine =< 1.5 x upper limit of normal (ULN); Note: if serum creatinine is > 1.5 x ULN, subject is eligible if the calculated creatinine clearance (CLcr) is >= 50 mL/min
* Total bilirubin =< 1.5 x ULN
* For patients without documented bone metastases or for patients with liver metastases: transaminases (aspartate aminotransferase [AST]/serum glutamic oxaloacetic transaminase [SGOT] and/or alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase [SGPT]) may be up to 2.5 x institutional ULN if alkaline phosphatase is =< ULN, or alkaline phosphatase may be up to 4 x ULN if transaminases are =< ULN
* For patients with documented bone metastases, the transaminases (AST/SGOT and/or ALT/SGPT) should be less than 2.5 x institutional ULN, without regard to the alkaline phosphatase level
* Sexually active males must use measures to prevent pregnancy in their partners while on STA-9090
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Major surgery within 4 weeks prior to first dose of STA-9090
* Poor venous access for study drug administration or would require a peripheral or central indwelling catheter for study drug administration; study drug administration via indwelling catheters is prohibited at this time
* Use of any chemotherapy or other standard systemic treatments for prostate cancer, including investigational agents within 2 weeks or 6 half- lives of the agent, whichever is shorter, prior to receiving STA-9090; there must be at least 2 weeks between the end of palliative radiation and the start of study drug and all radiation therapy (XRT)-associated toxicities resolved to Grade 1 or 0
* History of severe allergic or hypersensitivity reactions to excipients (e.g., Polyethylene glycol [PEG] 300 and Polysorbate 80 [i.e. docetaxel])
* Baseline QTc > 450 msec or previous history of QT prolongation while taking other medications
* Ventricular ejection fraction (Ef) =< 55% at baseline
* Any history of current coronary artery disease, myocardial infarction, angina pectoris, angioplasty or coronary bypass surgery
* History of current uncontrolled dysrhythmias, or requirement for antiarrhythmic medications, or Grade 2 or greater left bundle branch block
* New York Heart Association class II/III/IV congestive heart failure with a history of dyspnea, orthopnea, or edema that requires current treatment with angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, beta-blockers or diuretics
* Current or prior radiation therapy to the left hemithorax
* Treatment with chronic immunosuppressants (e.g. cyclosporine following transplantation)
* Uncontrolled intercurrent illness including, but not limited to, human immunodeficiency virus (HIV)-positive subjects receiving combination antiretroviral therapy, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, ventricular arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Other medications, or severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Heath, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (4):
- United States (4):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Medicine nd Denistry of New Jersey, Piscataway, New Jersey
  - University of Wisconsin Cancer Center Riverview, Wisconsin Rapids, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Started | 18
Completed | 17
Not Completed | 1
Not completed — Never rec'd treatment, but registered. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 68 [51 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: PFS Proportion Achieved With STA-9090 in Men With CRPC Who Have Received Prior Docetaxel Based Therapy
Description: Our primary objective was to determine the 6-month PFS rate by using a binary (yes/no) endpoint of 6 months of PFS. Treatment success was defined as achievement of at least 6 months of PFS. Patients who did not complete 6 months of ganetespib therapy for any reason (including death from any cause) were considered treatment failures and were recorded as not achieving the primary endpoint.
Time Frame: At 6 months
Measure: Number (90% Confidence Interval); unit: proportion with 6+ months PFS
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 18
proportion with 6+ months PFS | 0.0 [0.0 to 0.137]

2. Secondary Outcome: Percentage Change in PSA
Description: Percentage change in PSA from baseline.
Time Frame: From baseline to 12 weeks
Measure: Median (Full Range); unit: percentage change from baseline PSA
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 18
percentage change from baseline PSA | 78.65 [34.11 to 353.45]

3. Secondary Outcome: Overall Safety and Tolerability of STA-9090
Description: Overall safety and tolerability of STA-9090 by total number of grade 3 adverse events
Time Frame: Day 1, 8, and 15 of each course and at end of treatment
Measure: Number; unit: events of grade 3+ toxicity
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 18
events of grade 3+ toxicity | 35

4. Secondary Outcome: OS in Metastatic CRPC Who Have Received Prior Docetaxel Therapy
Description: Overall Survival (OS) in metastatic Castrate Resistant Prostate Cancer (CRPC) who have received prior docetaxel therapy using Kaplan-Meier method
Time Frame: From first dose to death or the date last known alive
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 18
months | 12.5 [1.5 to 17.7]

5. Secondary Outcome: Association of PFS With PSA
Description: Association of PFS with PSA using Cox PH regression model
Time Frame: At 6 months
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 18
Hazard Ratio | 1.000 [0.999 to 1.001]

6. Secondary Outcome: Potential Markers for Predicting Drug Response or Efficacy
Description: Potential markers for predicting drug response or efficacy : This is not a measurable outcome, but a possible entity for further study.
Time Frame: At baseline, day 1 of course 3, and end of treatment
Population: No data was collected for this outcome.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Serious Adverse Events (participants affected / at risk) | 10/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=18)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Alkaline phosphatase increased (Investigations) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Investigations, other (Investigations) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=18)
Alkaline phosphatase increased (Investigations) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Aspartate aminotransferase increase (Investigations) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 10 (10)
Fatigue (General disorders) | 7 (7)
Hematuria (Renal and urinary disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (8)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (7)
Lymphocyte count decreased (Investigations) | 7 (7)
Nausea (Gastrointestinal disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 9 (9)
Urinary tract infection (Infections and infestations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight loss (Investigations) | 5 (5)
White blood cell decreased (Investigations) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Pain (General disorders) | 3 (3)
Pain in extremity (General disorders) | 4 (4)
Serum amylase increased (Investigations) | 2 (2)
Infusion related reaction (General disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Alanine aminotransferase increased (Investigations) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (5)
Investigations - other (Investigations) | 2 (2)
Lipase increased (Investigations) | 3 (3)
Non-cardiac chest pain (General disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes